CLINICAL TRIAL: NCT03481842
Title: Safety, Tolerability and Efficacy of Vaginal Suppositories for Treatment of the Endometriosis
Acronym: ELTA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in study design and sponsor
Sponsor: BioGene Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C99884.337/18
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Endometriosis; Endometriosis Ovary; Endometriosis Externa; Endometriosis, Rectum
Keywords: Endometriosis; VEGF(R)
MeSH Terms: conditions — Endometriosis | interventions — linifanib; Afatinib; Axitinib

STUDY DESIGN:
Intervention Model Description: Single application in the morning of a vaginal suppository ELTA:
  Five days per week (with a treatment-free interval of two days in a row.) e.g. Monday and Tuesday - treatment-free days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaginal Suppositories (Experimental): Daily single administration of vaginal suppository in diagnosed endometriosis. Duration of admission-five days, two days-off. The total duration of treatment is 6 weeks. General course -30 vaginal suppositories ELTA
  The composition of the suppository:
  * Axitinib (inhibitor of VEGFR1, VEGFR2, VEGFR3, PDGFRβ and c-Kit) in a minimally sufficient therapeutic dose
  * Afatinib (BIBW2992) EGFR / HER2 including EGFR (wt), EGFR (L858R), EGFR (L858R / T790M) and HER2 inhibitor - minimally sufficient therapeutic dose
  * Linifanib (ABT-869) ATP-competitive VEGFR / PDGFR inhibitor for KDR, CSF-1R, Flt-1/3 and PDGFRβ - minimally sufficient therapeutic dose
  Interventions: Biological: Linifanib; Drug: BIBW2992; Drug: Axitinib

INTERVENTIONS:
Biological: Linifanib — in a minimally sufficient therapeutic dose
  Other Names: ABT869
Drug: BIBW2992 — in a minimally sufficient therapeutic dose
  Other Names: Afatinib; Giotrif
Drug: Axitinib — in a minimally sufficient therapeutic dose
  Other Names: AG013736;; Inlyta

SUMMARY:
Background:

Endometriosis is a chronic gynecological disease with the growth of endometrial tissue outside the endometrium. In all its properties, this tissue is similar to the mucous membrane of the uterus.

Types of endometriosis:

Endometriosis is divided into genital and extragenital. Genital endometriosis is internal and external. When the inner is affected by the uterus, with the external - the ovaries, tubes, vagina and external genital organs are affected. Extragenital endometriosis can affect various organs of the abdominal cavity.

Drug treatment does not show high effectiveness. Surgery / laparoscopic is currently considered the gold standard treatment for this problem, including infertility treatment.

The purpose of our studies is to achieve substantial results with respect to tolerability, safety and clinical efficacy of vaginal suppository ELTA for treatment of the endometriosis.

Methods:

Phase I clinical trial to be conducted at Cancer Center to hold under the aegis UniversitätsSpital Zürich from May 2018 to September 2018.

Ninety-four patients with the form of genital endometriosis will take part in the studies. The study was approved by the Ethics Committee at the Cancer Institute no C99884.01FH339

DETAILED DESCRIPTION:
The composition of the endometrium includes epithelial cell layers lining the uterine cavity, and deeper stroma, including the secretory glands. Each layer is characterized by the presence of a large number of blood vessels, through which a sufficient amount of blood is delivered. A large number of these vessels and arteries go to the surface layers due to myometrium and form a capillary network in the stroma.

In the vaginal suppositories, the investigators applied minimally therapeutic doses of inhibitors of neoangiogenesis, as well as other components that caused the pathological growth of the endometrium.

Anti-angiogenic therapy - inhibition of proliferative processes in the vascular wall of capillaries and small vessels in the endometrium, is the determining factor of the therapeutic effect of endometriosis when treated with vaginal suppositories.

The composition of the suppository:

* Axitinib, Afatinib, Linifanib (ABT-869) in a minimally sufficient therapeutic doses
* Auxiliary substances that ensure a uniform release of active components from suppositories, taking into account the dependence of this process on the chemical nature of the basis, surfactant, dissolution medium.

(the composition and amount of excipients are maximally optimal for bioavailability of drugs from suppositories, taking into account the pharmacokinetics, pharmacodynamics and synergy of active drugs) This therapy has a slight teratogenic effect, which should be taken into account when planning pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* verification of endometriosis
* signed agreement of informed consent
* agreement with information on the nature, relevance and scope of the investigation, as well as the expected results and undesirable consequences of IMD

Exclusion Criteria:

* use of not permitted contraception or not willing to use contraception
* pregnancy or lactation
* planned pregnancy in the next 36 months with the consent to participate in that clinical trial
* use of any other intravaginal medicinal product or medical device
* known hypersensitivity to one or more of the active and / or inactive ingredients
* acute or chronic renal failure
* acute or chronic heart failure
* the patient's reluctance to follow the trial protocol
* chronic alcoholism
* drug addiction
* use of antidepressants (during participation in trial)

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Local tolerability of the vaginal suppository ELTA defined as a cumulative sum of clinical signs for each patient | 6 weeks
  Local tolerability of the vaginal suppositories ELTA will be defined as a cumulative sum score of the solicited local /vaginal (consisting of subjectively experienced symptoms rated by the patient: burning, itching, bleeding, pain, dryness and objectively documented findings rated by the physician: redness, petechial bleeding, dryness, swelling) for each patient after every weeks of application (scored from 0 [none/normal] to 5 [severe]) Weekly visit of patients every seventh day from the beginning of treatment.
  SCALE EVALUATION EVENTS
  * burning - 2 points,
  * dryness - 1 point,
  * painful symptom- 3 points,
  * itching - 1 point,
  * bleeding - 5 points,
  If there is bleeding or the development of edema - the study for the patient will be stopped.

SECONDARY OUTCOMES:
Subjective symptoms (local tolerability) | 7 weeks
  Each of the subjective symptoms (scored from 0 [none/normal] to 5 [severe]) from the first visit (after the first application)/ A detailed description of the symptoms in each visit (with endoscopic photofixation of the endometriosis surface)

OTHER OUTCOMES:
Objective findings | 7 weeks
  Each of the objective symptoms (scored from 0 [none/normal] to 3 [severe]) from the first visit (after the first application).
  * dryness, itching, hyperemia of the perineum - 1 point,
  * pain syndrome with itching / dryness or without - 2 points,
  * bleeding with pain syndrome (or other symptoms / without them - 3 points,
  A detailed description of the symptoms in each visit (with endoscopic photofixation of the endometriosis surface)
Global judgement of tolerability | 4 weeks
  Global judgement of tolerability by investigator and patients. The scores of the Clinical Global Impression (CGI) Scale.
Safety evaluation of therapy | 15 weeks
  Safety evaluation of therapy. Drugs safety will be evaluated by assessment of adverse events ( ADRs).
Serious Adverse Event. | up to 15 weeks
  Occurrence of AE / SAE / ADE / SADE. Characteristics of occured AE / SAE / ADE / SADE
Change in pH-value from vaginal smear | up to 6 weeks
  pH-value from vaginal smear at every visit for each patient after the 3rd and 6th week of application of suppositories.
Change in Vaginal flora | up to 15 weeks
  Vaginal flora (Lactobacillus spp., Atopobium vaginae and Gardnerella vaginalis) on the first day of intake (before using the first suppository) and on the day of termination of therapy
Other signs of assessing the hip therapy | up to 15 weeks
  Mandatory Clinical blood test for each patient after the 3rd and 6th week of application of suppositories.
  A control blood test on the first day of the 15th week after the start of the first suppository

CONTACTS AND LOCATIONS:
Locations (1):
- BioGene Pharmaceutical Ltd., Basel, Вâlе, Switzerland